CLINICAL TRIAL: NCT00043069
Title: Osteoporosis Prevention in Prostate Cancer Patients Receiving Androgen Ablation Therapy: A Phase III Randomized, Placebo-Controlled, Double-Blind Study
Brief Title: Calcium With or Without Estrogen and/or Risedronate in Preventing Osteoporosis in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N01C8; NCI-2012-02482 (Registry Identifier: CTRP (Clinical Trials Reporting System)); NCI-P02-0229; CDR0000069502 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Osteoporosis; Prostate Cancer
Keywords: osteoporosis; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Osteoporosis; Prostatic Neoplasms | interventions — Calcium Carbonate; Cholecalciferol; Estrogen Antagonists; Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I: calcium + cholecalciferol + placebo + estrogen (Active Comparator): Patients receive oral calcium, oral cholecalciferol, oral risedronate placebo, and oral estrogen placebo daily.
  Treatment in all arms continues for 2 years.
  Quality of life is assessed at baseline, monthly for 6 months, and then at 1 and 2 years.
  Bone mineral density is assessed at baseline, 6 months, and 1 and 2 years.
  Interventions: Dietary Supplement: calcium carbonate; Dietary Supplement: cholecalciferol; Drug: Estrogen Antagonists; Other: placebo
- Arm II: calcium + cholecalciferol + risedronate + estrogen (Experimental): Patients receive oral calcium, oral cholecalciferol, oral risedronate, and oral estrogen placebo daily.
  Treatment in all arms continues for 2 years.
  Quality of life is assessed at baseline, monthly for 6 months, and then at 1 and 2 years.
  Bone mineral density is assessed at baseline, 6 months, and 1 and 2 years.
  Interventions: Dietary Supplement: calcium carbonate; Dietary Supplement: cholecalciferol; Drug: Estrogen Antagonists; Drug: risedronate sodium
- Arm III: calcium + cholecalciferol + placebo + estrogen (Placebo Comparator): Patients receive oral calcium, oral cholecalciferol, low-dose oral conjugated estrogens, and oral risedronate placebo daily.
  Treatment in all arms continues for 2 years.
  Quality of life is assessed at baseline, monthly for 6 months, and then at 1 and 2 years.
  Bone mineral density is assessed at baseline, 6 months, and 1 and 2 years.
  Interventions: Dietary Supplement: calcium carbonate; Dietary Supplement: cholecalciferol; Drug: Estrogen Antagonists; Other: placebo
- Arm IV: calcium + cholecalciferol + risedronate + estrogen (Experimental): Patients receive oral calcium, oral cholecalciferol, low-dose oral conjugated estrogens, and oral risedronate daily.
  Treatment in all arms continues for 2 years.
  Quality of life is assessed at baseline, monthly for 6 months, and then at 1 and 2 years.
  Bone mineral density is assessed at baseline, 6 months, and 1 and 2 years.
  Interventions: Dietary Supplement: calcium carbonate; Dietary Supplement: cholecalciferol; Drug: Estrogen Antagonists; Drug: risedronate sodium

INTERVENTIONS:
Dietary Supplement: calcium carbonate
Dietary Supplement: cholecalciferol
Drug: Estrogen Antagonists
Drug: risedronate sodium
  Arms: Arm II: calcium + cholecalciferol + risedronate + estrogen; Arm IV: calcium + cholecalciferol + risedronate + estrogen
Other: placebo
  Arms: Arm I: calcium + cholecalciferol + placebo + estrogen; Arm III: calcium + cholecalciferol + placebo + estrogen

SUMMARY:
RATIONALE: Preventing bone loss in patients who are undergoing androgen ablation for prostate cancer may decrease the risk of fractures and may help patients live more comfortably. It is not yet known whether calcium is more effective with or without estrogen and/or risedronate in preventing osteoporosis.

PURPOSE: Randomized phase III trial to compare the effectiveness of two forms of calcium with or without estrogen and/or risedronate in preventing osteoporosis in patients with prostate cancer who are receiving androgen ablation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the change in bone mineral density in patients with prostate cancer who are receiving androgen-ablation therapy treated with calcium and cholecalciferol with or without conjugated estrogens and with or without risedronate.
* Compare the toxicity of these regimens in these patients.
* Compare the changes in bone markers in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare hot flashes in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to duration of therapy with luteinizing hormone-releasing hormone agonists (no more than 30 days vs 31 to 150 days vs 151 to 365 days vs more than 365 days). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral calcium, oral cholecalciferol, oral risedronate placebo, and oral estrogen placebo daily.
* Arm II: Patients receive oral calcium, oral cholecalciferol, oral risedronate, and oral estrogen placebo daily.
* Arm III: Patients receive oral calcium, oral cholecalciferol, low-dose oral conjugated estrogens, and oral risedronate placebo daily.
* Arm IV: Patients receive oral calcium, oral cholecalciferol, low-dose oral conjugated estrogens, and oral risedronate daily.

Treatment in all arms continues for 2 years.

Quality of life is assessed at baseline, monthly for 6 months, and then at 1 and 2 years.

Bone mineral density is assessed at baseline, 6 months, and 1 and 2 years.

PROJECTED ACCRUAL: A total of 282 patients (70 per treatment arm) will be accrued for this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of prostate cancer

  * No evidence of metastatic bony disease* NOTE: *Elevated prostate-specific antigen (PSA) allowed
* Meets one of the following criteria:

  * Currently on treatment with androgen-ablation therapy in the adjuvant setting
  * Rising PSA without other evidence of recurrent disease with planned treatment for at least 6 months
* No known osteoporosis or prior osteoporotic fracture

  * Osteoporosis defined as bone density at the hip or spine of more than 2.5 standard deviations below the mean for young men

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* SGOT or SGPT no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase normal OR no greater than 1.5 times ULN with a normal bone scan

Renal

* Creatinine no greater than 1.5 times ULN
* No prior symptomatic hypercalcemia or hypocalcemia

Cardiovascular

* No active heart disease
* No congestive heart failure under active treatment
* No myocardial infarction within the past 5 years
* No coronary artery disease (CAD) with recent myocardial infarction

  * Patients with a remote history of CAD who are only on medical treatment (e.g., antilipid agents) are allowed
* No prior thrombosis (deep vein thrombosis, stroke, or pulmonary embolism) or other known hypercoagulable state other than cancer

Other

* Fertile patients must use effective contraception
* Triglycerides no greater than 250 mg/dL (treatment allowed)
* Able to complete questionnaire(s) by self or with assistance
* Able to swallow pills
* No prior hyperlipidemia (e.g., prior familial hyperlipidemia or fasting triglyceride greater than 250 mg/dL within the past 6 months)
* No sarcoidosis
* No parathyroid dysfunction
* No intolerance to bisphosphonates

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent systemic steroids

Radiotherapy

* No concurrent radiotherapy

Surgery

* More than 3 months since prior and no concurrent dental extraction, root canal, or dental implantation

Other

* No prior bisphosphonates
* More than 5 years since prior percutaneous transluminal coronary angioplasty

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2002-11; Primary Completion 2006-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density by test at 1 and 2 years | Up to 2 years

SECONDARY OUTCOMES:
Toxicity questionnaires every 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (114):
- United States (112):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Alegent Health Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Cancer Center at Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Brainerd Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Mercy and Unity Hospitals, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Cancer Center at Creighton University Medical Center, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Health System, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
- Canada (2):
  - Pasqua Hospital, Regina, Saskatchewan
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Result] Kearns AE, Northfelt DW, Dueck AC, Atherton PJ, Dakhil SR, Rowland KM Jr, Fuloria J, Flynn PJ, Dentchev T, Loprinzi CL. Osteoporosis prevention in prostate cancer patients receiving androgen ablation therapy: placebo-controlled double-blind study of estradiol and risedronate: N01C8. Support Care Cancer. 2010 Mar;18(3):321-8. doi: 10.1007/s00520-009-0655-x. Epub 2009 May 27. PMID 19468757